CLINICAL TRIAL: NCT03700892
Title: In-vivo Effects of E-cigarette Aerosol on Innate Lung Host Defense
Acronym: Cinimic
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19 has been shown to increase risk associated with vaping. To increase participant safety and use real world vaping habits, the investigators plan to continue studying vaping effects on the airways in an observational format.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 17-2275; R01HL139369 (NIH)
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Results first posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-03

CONDITIONS: Smoking; Healthy
Keywords: e-cig; E-cigarette; Electronic cigarette; Vaping
MeSH Terms: conditions — Smoking; Vaping

STUDY DESIGN:
Intervention Model Description: Controls will not be randomized and will not receive the study intervention.
Who Masked: Participant, Outcomes Assessor
Masking Description: The e-liquids will be maintained by an individual not active in the study procedures or analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cinnamaldehyde, then PG/VG (Experimental): Participants will inhale cinnamaldehyde e-liquid in 6, 5-minute paced vaping segments (1 puff/minute) over 1 hour. A 2-3 week washout period will follow. Then participants will inhale Propylene Glycol/Vegetable Glycerin (PG/VG) e-liquid in 6, 5-minute paced vaping segments (1 puff/minute) over 1 hour.
  Interventions: Other: Cinnamaldehyde e-liquid; Other: PG/VG e-liquid
- PG/VG, then Cinnamaldehyde (Experimental): Participants will inhale PG/VG e-liquid in 6, 5-minute paced vaping segments (1 puff/minute) over 1 hour. A 2-3 week washout period will follow. Then participants will inhale cinnamaldehyde e-liquid in 6, 5-minute vaping segments (1 puff/minute) over 1 hour.
  Interventions: Other: Cinnamaldehyde e-liquid; Other: PG/VG e-liquid
- Healthy Controls (No Intervention): Participants will only undergo the baseline testing and thus serve as a non-exposed/non-vaping control group.

INTERVENTIONS:
Other: Cinnamaldehyde e-liquid — Participants will inhale an e-liquid that contains cinnamaldehyde from Vapor Shark DNA 250™ e-cigarette device allowing manual control and vapor setting recordings (voltage, wattage, puff volume, and frequency).
  Other Names: Cinnamon
  Arms: Cinnamaldehyde, then PG/VG; PG/VG, then Cinnamaldehyde
Other: PG/VG e-liquid — Participants will inhale an e-liquid that contains PG/VG from the Vapor Shark DNA 250™ e-cigarette device allowing manual control and vapor setting recordings (voltage, wattage, puff volume, and frequency).
  Other Names: Placebo
  Arms: Cinnamaldehyde, then PG/VG; PG/VG, then Cinnamaldehyde

SUMMARY:
While e-cigs are commonly represented as safer alternatives to tobacco cigarettes, little is known regarding the health effects of their short- or long-term use. The responses and the e-cig components exerting these effects on the airways are largely unknown. This study will identify if specific e-cig flavors modify respiratory immune responses. This study will determine the effects of cinnamaldehyde (CA)-containing e-cigarettes on airway epithelial cell ciliary function (i.e., MCC) in humans. Additionally the study will determine the effects of CA-containing e-cigarettes on airway immune cells obtained through induced sputum (SI) after inhalation of CA-containing e-cig aerosols to determine CA-induced effects on a) immune cell function (e.g., phagocytosis, respiratory burst), b) immune cell surface phenotype, and c) mediator production in humans in vivo.

DETAILED DESCRIPTION:
Investigators will evaluate the acute effect of CA-flavored e-cigs on MCC and IS immune cells in up to 32 healthy, young adults who are current e-cig users with a total of less than 10 pack-years cigarette smoking history. MCC will be measured by gamma scintigraphy at baseline and following controlled vaping of e-liquids with and without cinnamon flavoring. Two different e-liquids (one completely devoid and one containing at least 30 mM CA similar to "Hot Cinnamon Candies" which is commercially available) will be used for two separate randomized vaping sessions.

The randomization scheme for the two different e-liquids (e-liquids with and without CA) will be generated by using the Web site Randomization.com (http://www.randomization.com), assigned treatment Regimen A and B by an assigned study team member, and provided to the study team. This individual will also be responsible for loading the e-cigarette with the appropriate solution for that session prior to the vaping sessions.

Participants will undergo baseline testing during the screening visit, which will occur 2-3 weeks prior to the first controlled vaping session. Investigators will also recruit non-vaping control subjects (n=32), who will only undergo the baseline testing and thus serve as a non-exposed/non-vaping control group. will aim to recruit similar numbers of males and females in both cohorts. While investigators cannot guarantee age-matching and sex-matching in these cohorts, based on our previous studies, investigators do not expect to find significant age and sex differences in the two cohort. In addition, potential confounders, such as age, sex, and BMI will be included as covariates in our multivariate analysis.

Observations obtained from the non-vaping control group will provide necessary information on potential baseline differences in the two cohorts (i.e. current vapers versus non-vaping controls). These data from the non-vaping control group are important to provide a reference for any potential CA-induced changes in the vaping group. Hence, there are two stages of the study:

Stage 1. A cross sectional observational cohort comparison of baseline MCC and IS immune cells in a reference cohort of n=32 non-vaping control subjects and E-cig cohort of n=32 currently vaping subjects (confounding based on other variables such as BMI, sex, age is possible for this stage).

Stage 2. A randomized comparison of changes in MCC and IS immune cells after Regimen A (e-cig us without CA) and Regimen B (e-cig use with CA). The cohort of e-cig users will undergo a randomized 2-treatment, 2-period, 2-sequence crossover study of CA exposure.

For stage 1, baseline measurements of Tc99m-SC clearance will be used to measure each subject's normal baseline MCC and IS immune cell characteristics. For both stages, subjects will be asked to complete a vaping diary to record information on the device and e-liquids (name/vendor/e-liquids/puffs/device settings) used during their normal vaping sessions for the entire duration of the study. In addition, for stage 2, participants will be asked to maintain their current habits for the duration of the study, not to significantly increase or decrease their vaping patterns, including the nicotine concentrations of their e-liquids.

For stage 2, for each e-cig vaping session (Training and MCC Test Days), subjects will be asked to follow a laboratory-based protocol involving 6, 5-minute paced vaping segments (1 puff/minute) over a 1 hour time period, vaping the e-liquid with and without CA provided by us. On each Test Day, participants will undergo the vaping protocol immediately prior to inhalation of the Tc99m-SC (10 min between end of vaping and inhalation of Tc99m-SC). An initial deposition scan of Tc99m-SC will then be obtained followed by dynamic imaging of the lung with subjects seated in front of the gamma camera to determine potential changes in MCC induced by acute exposure to CA-flavored e- cigarettes. Induced sputum samples will be collected at baseline, and after each MCC scan.

24 hours after completion of the MCC scans. The two randomized vaping sessions will be separated by 2-3 weeks. While there are no data providing specific information on the duration needed to washout the effects of CA on MCC, previous studies examining changes in MCC following inhalation of other aerosols have shown that this washout period is sufficient to prevent potential carryover between the two treatments.

ELIGIBILITY:
Inclusion Criteria:

* An equal number of participants who currently use a vaping device and those who do not use a vaping device
* Age 18-40
* Must have a Forced Vital Capacity (FVC) and Forced Expiratory Volume in 1 second (FEV₁) of at least 80% of predicted. Participants who fall out of the normal range will be offered a copy of the test to share with their personal physician.

Exclusion Criteria:

* Any pre-existing lung disease (asthma, cystic fibrosis, etc.)
* Any significant chronic illness, such as, but not limited to, heart disease, uncontrolled hypertension, diabetes, auto-immune disease
* Any use of tobacco products (other than e-cig) in the past 3 months, or a greater than 10 pack year history of smoking cigarettes
* Pregnant or nursing women
* Participants with a history of radiation exposure in the past year which exceeds annual safe limits.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ilona Jaspers, PhD, Principal Investigator — University of North Carolina
Locations (1):
- UNC Center for Environmental Medicine, Asthma and Lung Biology, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, ﬁgures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.
  Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata
  Requests for access to individual participant data should be sent to bring44@email.unc.edu or carole.robinette@med.unc.edu. Access will be granted after a data access agreement has been signed with UNC.

REFERENCES:
- [Derived] Bennett WD, Clapp PW, Zeman KL, Wu J, Ring B, Jaspers I. Acute Effect of E-Cigarette Inhalation on Mucociliary Clearance in E-Cigarette Users. J Aerosol Med Pulm Drug Deliv. 2024 Aug;37(4):167-170. doi: 10.1089/jamp.2023.0027. Epub 2024 Apr 22. PMID 38687136

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After qualifying, all participants move to the baseline day in which an mucociliary clearance (MCC) scan and sputum are collected for baseline measurements. The vaping participants continue on to the crossover design for CA and PG/VG sessions followed by MCC scans and sputum collections for post exposure measurements.
Groups:
- Cinnamaldehyde, Then PG/VG: Participants will inhale cinnamaldehyde(CA) e-liquid in 6, 5-minute paced vaping segments (1 puff/minute) over 1 hour. A 2-3 week washout period will follow. Then participants will inhale Propylene Glycol/Vegetable Glycerin (PG/VG) e-liquid in 6, 5-minute paced vaping segments (1 puff/minute) over 1 hour.
  Cinnamaldehyde e-liquid: Participants will inhale an e-liquid that contains cinnamaldehyde from Vapor Shark DNA 250™ e-cigarette device allowing manual control and vapor setting recordings (voltage, wattage, puff volume, and frequency).
  PG/VG e-liquid: Participants will inhale an e-liquid that contains PG/VG from the Vapor Shark DNA 250™ e-cigarette device allowing manual control and vapor setting recordings (voltage, wattage, puff volume, and frequency).
Period: Baseline
Arm/Group | Cinnamaldehyde, Then PG/VG | PG/VG, Then Cinnamaldehyde | Healthy Controls
Started | 15 | 0 | 4
Completed | 15 | 0 | 4
Not Completed | 0 | 0 | 0
Period: First Intervention (Single 1-Day Visit)
Arm/Group | Cinnamaldehyde, Then PG/VG | PG/VG, Then Cinnamaldehyde | Healthy Controls
Started | 1 | 4 | 0
Completed | 1 | 4 | 0
Not Completed | 0 | 0 | 0
Period: Washout (2-3 Weeks)
Arm/Group | Cinnamaldehyde, Then PG/VG | PG/VG, Then Cinnamaldehyde | Healthy Controls
Started | 1 | 4 | 0
Completed | 1 | 4 | 0
Not Completed | 0 | 0 | 0
Period: Second Intervention (Single 1-Day Visit)
Arm/Group | Cinnamaldehyde, Then PG/VG | PG/VG, Then Cinnamaldehyde | Healthy Controls
Started | 1 | 4 | 0
Received Intervention | 1 | 3 | 0
Completed | 1 | 3 | 0
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Treated Participants: All participants inhaled cinnamaldehyde e-liquid or Propylene Glycol/Vegetable Glycerin (PG/VG) e-liquid in either Period 1 or Period 2 as per randomization schedule.
  Cinnamaldehyde e-liquid: Participants will inhale an e-liquid that contains cinnamaldehyde from Vapor Shark DNA 250™ e-cigarette device allowing manual control and vapor setting recordings (voltage, wattage, puff volume, and frequency).
  PG/VG e-liquid: Participants will inhale an e-liquid that contains PG/VG from the Vapor Shark DNA 250™ e-cigarette device allowing manual control and vapor setting recordings (voltage, wattage, puff volume, and frequency).
- Total: Total of all reporting groups
Arm/Group | All Treated Participants | Healthy Controls | Total
Number analyzed (Participants) | 15 | 4 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 4 | 19
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 12 | 1 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 13 | 4 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 11 | 4 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 4 | 19

OUTCOME MEASURES:

1. Primary Outcome: CA-induced Changes in Whole Lung MCC
Description: Absolute values of whole lung MCC at baseline compared to after CA vaping session. Absolute repeat values of Whole lung MCC = average % mucus cleared from the whole lung over a 90-minute period.
Time Frame: Through study completion, an average of three months
Population: The healthy control participants only undergo the baseline testing and thus serve as a non-exposed/non-vaping control group. This Primary outcome does not apply to the healthy control group as they did not receive the intervention and only baseline data was collected.
Measure: Mean (Standard Deviation); unit: percent clearance
Groups:
- Cinnamaldehyde: Participants will inhale cinnamaldehyde e-liquid in 6, 5-minute paced vaping segments (1 puff/minute) over 1 hour. A 2-3 week washout period will follow.
  Cinnamaldehyde e-liquid: Participants will inhale an e-liquid that contains cinnamaldehyde from Vapor Shark DNA 250™ e-cigarette device allowing manual control and vapor setting recordings (voltage, wattage, puff volume, and frequency).
- PG/VG: Participants will inhale PG/VG e-liquid in 6, 5-minute paced vaping segments (1 puff/minute) over 1 hour. A 2-3 week washout period will follow.
  PG/VG e-liquid: Participants will inhale an e-liquid that contains PG/VG from the Vapor Shark DNA 250™ e-cigarette device allowing manual control and vapor setting recordings (voltage, wattage, puff volume, and frequency).
Arm/Group | Cinnamaldehyde | PG/VG
Number analyzed (Participants) | 4 | 5
percent clearance | 41 (5) | 27 (17)

2. Secondary Outcome: CA-induced Changes in Regional Lung MCC
Description: Absolute repeat values of Central and Peripheral lung MCC = average % mucus cleared from the Central and Peripheral lung over a 90-minute period. This will assess clearance rates from the central (C) and peripheral (P) regions as secondary endpoints that may reflect differential effects between a region with relatively more (C) vs. less (P) large bronchial airways.
Time Frame: Through study completion, an average of three months
Measure: Mean (Standard Deviation); unit: percent clearance
Arm/Group | Cinnamaldehyde | PG/VG
Number analyzed (Participants) | 4 | 5
percent clearance
  Central Lung | 43 (12) | 25 (32)
  Peripheral Lung | 33 (3) | 24 (6)

3. Secondary Outcome: Percent Polymorphonuclear Leukocytes (PMN) in Induced Sputum
Description: Percent change of PMNs in vapers from baseline compared to post CA vaping session. Percent change in PMNs in vapers from baseline compared to post PG/VG vaping session are included as an additional comparison.
Time Frame: Through study completion, an average of three months
Population: The healthy control participants only undergo the baseline testing and thus serve as a non-exposed/non-vaping control group. This outcome does not apply to the healthy control group as they did not receive the intervention and only baseline data was collected.
Measure: Mean (Standard Error); unit: percent PMN
Arm/Group | Cinnamaldehyde | PG/VG
Number analyzed (Participants) | 4 | 5
percent PMN | 3.6 (7.2) | 89.4 (5.8)

4. Secondary Outcome: Absolute Values of Whole Lung MCC for Each Group
Description: Baseline Differences in Whole lung MCC clearance rates in Non-smokers/Non-vapers as Compared to E-cigarette Users. Absolute group values of Whole Lung MCC =average % mucus cleared from the whole lung over a 90-minute period.
Time Frame: Start of study, up to three months
Population: Includes all participants who completed the baseline MCC scan.
Measure: Mean (Standard Deviation); unit: percent clearance
Groups:
- E-cigarette Users: Baseline MCC scans and sputum collection performed prior to randomization.
- Non-smoker/Non-vaper Healthy Controls: Baseline MCC scans and sputum collection.
Arm/Group | E-cigarette Users | Non-smoker/Non-vaper Healthy Controls
Number analyzed (Participants) | 15 | 4
percent clearance | 17 (8) | 14 (6)

5. Other Pre Specified Outcome: CA-Induced Changes in Immune Cell Function
Description: Percent change from baseline in phagocytosis
Time Frame: Through study completion, an average of three months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Peripheral Blood Mononuclear Cell Analysis
Description: Percent change in cell counts as compared to baseline
Time Frame: Through study completion, an average of three months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Blood Serum Analysis of Inflammatory Mediators
Description: Percent change of mediator expression as compared to baseline
Time Frame: Through study completion, an average of three months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: CA-Induced Changes in Epithelial Lining Fluid
Description: Pre-vaping session versus post-vaping session expressed as a percent change
Time Frame: Through study completion, an average of three months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: CA-Induced Changes in Epithelial Lining Fluid 24 Hours After Vaping Session
Description: Percent change as compared to post-vaping session sample
Time Frame: Through study completion, an average of three months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Changes in Epithelial Lining Fluid
Description: Percent change as compared to baseline
Time Frame: Through study completion, an average of three months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Tidal Volume Subjects Own E-cigarette Device
Description: Tidal Volume in milliliters
Time Frame: Through study completion, an average of three months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Respiratory Rate With Subjects Own E-cigarette Device
Description: Respiratory Rate in breaths per minute
Time Frame: Through study completion, an average of three months
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Minute Ventilation With Subjects Own E-cigarette Device
Description: Minute Ventilation in L/min
Time Frame: Through study completion, an average of three months
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Inspiratory Flow With Subjects Own E-cigarette Device
Description: Inspiratory flow in L/min
Time Frame: Through study completion, an average of three months
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Expiratory Flow With Subjects Own E-cigarette Device
Description: Expiratory flow in L/min
Time Frame: Through study completion, an average of three months
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Tidal Volume With Investigator E-cigarette Device
Description: Tidal Volume in milliliters
Time Frame: Through study completion, an average of three months
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Respiratory Rate With Investigator E-cigarette Device
Description: Respiratory Rate in breaths per minute
Time Frame: Through study completion, an average of three months
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Minute Ventilation With Investigator E-cigarette Device
Description: Minute Ventilation in L/min
Time Frame: Through study completion, an average of three months
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Inspiratory Flow With Investigator E-cigarette Device
Description: Inspiratory flow in L/min
Time Frame: Through study completion, an average of three months
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Expiratory Flow With Investigator E-cigarette Device
Description: Expiratory flow in L/min
Time Frame: Through study completion, an average of three months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the time a participant signed consent through completion of the second intervention, a total of up to 3 months.
Description: Adverse event data included all participants who received at least one dose of Cinnamaldehyde (CA) or Propylene Glycol/Vegetable Glycerin (PG/VG).
Groups:
- Cinnamaldehyde: Participants who inhaled cinnamaldehyde e-liquid in either Period 1 or Period 2 as per randomization schedule.
  Cinnamaldehyde e-liquid: Participants will inhale an e-liquid that contains cinnamaldehyde from Vapor Shark DNA 250™ e-cigarette device allowing manual control and vapor setting recordings (voltage, wattage, puff volume, and frequency).
- PG/VG: Participants who inhaled Propylene Glycol/Vegetable Glycerin (PG/VG) e-liquid in either Period 1 or Period 2 as per randomization schedule.
  PG/VG e-liquid: Participants will inhale an e-liquid that contains PG/VG from the Vapor Shark DNA 250™ e-cigarette device allowing manual control and vapor setting recordings (voltage, wattage, puff volume, and frequency).
Arm/Group | Cinnamaldehyde | PG/VG | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/92/NCT03700892/Prot_SAP_000.pdf